CLINICAL TRIAL: NCT06321159
Title: Investigation of the Effect of the Use of Mobile Software in Blood Pressure Management on the Quality of Life and Disease Self-Efficacy of Hypertensive Individuals Sheltered in Temporary Living Area
Brief Title: Investigation of the Effect of Mobile Software Use in Blood Pressure Management of Hypertensive Individuals on Quality of Life and Disease Self-Efficacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Fidan Balkaya, Research Asistant, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Nursing Dep.
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-03

CONDITIONS: Hypertension, Essential Hypertension
Keywords: Hypertension; Self-Efficacy; Quality of Life; Mobile Application
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Intervention Model Description: Our study has two groups of 78 participants each. Our study is an experimental study with pretest-posttest control group.
Who Masked: Participant
Masking Description: Participants will be determined blindly by being assigned by a site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): mobile application
  Interventions: Other: mobile application
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Other: mobile application — mobile application for diet, exercises and medication adherence
  Arms: Intervention Group

SUMMARY:
Hypertension is a prevalent health concern, affecting one in three adults globally, with the potential to lead to fatal complications. However, an alarming proportion of those diagnosed-four out of five individuals-struggle to effectively manage this condition. As such, the effective management of hypertension becomes paramount. A study conducted post-earthquake by a principal investigator and a scholarship recipient revealed that 47.9% of participants received a hypertension diagnosis, and a significant 67.8% ceased active management of the condition. Existing literature suggests a notable decline in the quality of life among individuals unable to manage hypertension effectively. While current research emphasizes the components of nutrition, exercise, and medication adherence in hypertension management, the integration of these components into mobile applications is notably lacking. This project seeks to enhance disease management for users by integrating crucial elements, including blood pressure measurement, into a user-friendly mobile application, thereby providing a distinctive contribution. The proposed application encompasses the recording of vital signs, integration of customized diet and exercise programs tailored for hypertension, and provision of consultancy services for identifying deviations in health status and implementing appropriate interventions. The integration of these components is anticipated to contribute to preventing or minimizing potential complications for the patient. Comprehensive studies incorporating such an approach are rarely encountered in the existing literature, enhancing the originality of this research. The projects overarching goal is to enable individuals to manage hypertension even in extraordinary circumstances, such as earthquakes. Consequently, the study will assess how the mobile application influences individuals; quality of life and disease self-efficacy.

Conducted between April 2024 and January 2026, the project adopts a pre-test post-test control group experimental design in the four most earthquake-affected provinces. It involves 614 individuals diagnosed with hypertension, residing in temporary living space in Malatya, Hatay, Kahramanmaraş, and Adıyaman, with 78, 77, and 74 participants in Malatya, Hatay, and Adıyaman, respectively. Data collection tools include the Personal Identification Information Form, Hypertension Self-Efficacy Scale, SF-36 Quality of Life Scale, and International Physical Activity Scale-Short Form, administered through face-to-face interviews. The mobile application development will be a collaborative effort with two faculty members from the Department of Computer Engineering and expert academicians. For the diet program within the application, eight questions will be used to uncover individuals' dietary preferences. Calculations based on Body Mass Index, basal metabolic rate, and daily energy requirements will inform the diet program, which will encompass five food groups and their caloric values. Notifications about diet adherence will be sent for each meal. In the exercise program, individuals will measure and record blood pressure and medication intake. Those with a blood pressure of 140/90 mmHg or higher will be included based on expert physician recommendations, with notifications for those exceeding 160/100 mmHg to consult a physician. A personalized exercise program will be created based on the OMRİ-RİS scale, supported by animations. Training videos for blood pressure measurements and medication adherence will be recorded and supervised by local academic nurse practitioners. Data analysis will utilize appropriate statistical tests conducted through computer programs. The project is anticipated to contribute significantly to researcher development, enhance quality of life and disease management, increase productivity, and establish new projects.

DETAILED DESCRIPTION:
Hypertension (HT) is a chronic disease that is widespread in the population and can lead to serious complications. Its high prevalence in Turkey and worldwide makes prevention and management of this disease critical. HT is a systemic disease characterised by persistently high blood pressure and is an important public health problem because it causes serious complications and is widely prevalent in the community (Hacıhasanoğlu Aşılar, 2015; Obesity, Dyslipidaemia, Hypertension Working Group, 2022). It is known that more than 30% of the adult population worldwide, i.e. more than one billion people worldwide, are affected by hypertension (PAHO, 2020). In our country, according to the data of the Turkish Society of Cardiology, the prevalence of hypertension in the adult population is 31.2% (Turkish Society of Cardiology, 2022). When hypertension is not well managed, it is known to be one of the leading causes of death leading to stroke and heart attack (Turkish Society of Cardiology, 2022; Zhang et al., 2021) and one of the most important risk factors for many chronic diseases such as diabetes and renal failure (Mancia et al., 2013). In a systematic review of the economic burden of cardiovascular disease and hypertension in low- and middle-income countries, it was found that the expenditures for hypertension and cardiovascular diseases in countries vary between 500 and 1500 dollars, and in countries such as Mexico, China, Brazil and India, it constitutes half of health expenditures (Gheorghe et al., 2018). Considering its prevalence in the world and in Turkey, and the high prevalence of material and moral damage, it becomes clear how important it is to prevent and manage hypertension. In recent studies, it has been found that individuals diagnosed with hypertension have a worse quality of life compared to those who do not have this diagnosis (Xu et al., 2016), and interventions for hypertension treatment and compliance positively affect the quality of life of individuals (Arija et al., 2018; Li et al., 2018; Souza et al., 2016; Zhang et al., 2021; Silva et al., 2020; Emre et al., 2020). (2018) examined the effect of physical activity on cardiovascular health, quality of life and blood pressure and found that physical activity increased the risk of cardiovascular disease by 1.19 points, quality of life by 4.45 to 14.62 points, and reduced systolic blood pressure by 8.68 mm Hg. In the meta-analysis study conducted by Souza and colleagues, it was found that training on hypertension management increased quality of life scores by an average of 8.26 (Souza et al., 2016). It has been reported that interventions for hypertension treatment and compliance positively affect the quality of life of individuals (Arija et al., 2018; Li et al., 2018; Souza et al., 2016; Zhang et al., 2021; Silva et al., 2020; Emre et al., 2020). Recent studies have addressed different aspects of hypertension such as quality of life, diet, exercise, and economic burden. However, it was observed that technology was not integrated in the management of hypertension in these studies.

It is seen that lifestyle changes such as nutrition and exercise are effective in both prevention and management of hypertension (Hacıhasanoğlu & Gözüm, 2011, Jones et al., 2020; Ozemek et al., 2018; Ventura & Lavia, 2018). Although excessive sodium intake among dietary factors predisposes individuals to the development of hypertension, dietary interventions for sodium restriction are still considered a popular recommendation for lowering blood pressure (Lackland et al., 2007; Whelton et al., 2018; World Health Organization, 2012). The Dietary Approaches to Stop Hypertension (DASH) diet and the Mediterranean diet are examples of effective dietary interventions to lower blood pressure based on healthy eating strategies. The DASH diet is a dietary model that emphasises the consumption of whole grain foods, legumes, oilseeds, fish and poultry, fruits, vegetables and low-fat dairy products, while restricting the consumption of red meat, high-fat and sugary foods and beverages. On the other hand, in this diet model, it was emphasised that the daily sodium intake of hypertensive individuals should be below 1500 mg (3.75 g salt) in order to reduce blood pressure (Filippou et al., 2020). In addition, it is seen that the content of the DASH diet is consistent with the nutritional recommendations of the World Health Organization, the American Heart Association and the Turkish Society of Hypertension and Kidney Diseases, which are effective in lowering blood pressure (). In the meta-analysis study conducted by Schwingshackl et al. (2019), it was revealed that the DASH diet reduced systolic blood pressure by 90% and diastolic blood pressure by 91%. In addition to reducing sodium intake, healthy dietary patterns with high potassium, calcium, magnesium and fibre content and low trans/saturated/total fat and dietary cholesterol content can also be considered as beneficial components of blood pressure. Indeed, recent findings have shown that the combination of low sodium and a healthy diet can lower blood pressure by approximately 50% more than low sodium intake alone (Filippou et al., 2022). In the literature, there are studies revealing that exercise has an effect on hypertension as well as dietary practices. It is seen that these exercises mostly consist of aerobic, resistance and combined exercise applications (Lopes et al., 2018, Pescatello, 2019). Regular aerobic exercise has been found to help reduce systolic and diastolic blood pressure by 8.3 and 5.2 mm Hg, respectively (Cornelissen & Smart, 2013). Aerobic exercise has also been found to have positive effects on pulse wave velocity, which is used as the gold standard in determining arterial stiffness (Zhang et al., 2018). In addition, it is seen that the content of the DASH diet is consistent with the nutritional recommendations of the World Health Organization, the American Heart Association and the Turkish Society of Hypertension and Kidney Diseases, which are effective in lowering blood pressure (). In the meta-analysis study conducted by Schwingshackl et al. (2019), it was revealed that the DASH diet reduced systolic blood pressure by 90% and diastolic blood pressure by 91%. In addition to reducing sodium intake, healthy dietary patterns with high potassium, calcium, magnesium and fibre content and low trans/saturated/total fat and dietary cholesterol content can also be considered as beneficial components of blood pressure. Indeed, recent findings have shown that the combination of low sodium and a healthy diet can lower blood pressure by approximately 50% more than low sodium intake alone (Filippou et al., 2022). In the literature, there are studies revealing that exercise has an effect on hypertension as well as dietary practices. It is seen that these exercises mostly consist of aerobic, resistance and combined exercise applications (Lopes et al., 2018, Pescatello, 2019). Regular aerobic exercise has been found to help reduce systolic and diastolic blood pressure by 8.3 and 5.2 mm Hg, respectively (Cornelissen & Smart, 2013). Aerobic exercise has also been found to have positive effects on pulse wave velocity, which is used as the gold standard in determining arterial stiffness (Zhang et al., 2018). Dynamic resistance exercises are also frequently performed in hypertensive individuals. The rationale for this is that during dynamic RE, blood flow is restricted during the contraction phase, but increases during the relaxation phase, resulting in more O2 delivery and oxidative metabolism (Williams et al., 2018). It is stated that there are positive effects on systolic and diastolic blood pressure after the application of resistance exercises with resistance tyres (Henkin et al., 2023). The use of resistance bands offers the opportunity for extremely safe and objective exercise practice. The intensity of the exercise can be determined by determining the degree of difficulty perceived by the practitioner. Therapeutic effect can be seen in hypertensive individuals with resistance exercises to be applied to major muscle groups. It has been stated that diaphragmatic breathing technique inhibits sympathetic nerve activities and chemoreflex activation by activating pulmonary-cardiac mechanoreceptors and thus helps arteriolar dilatation (Wang et al., 2010; Yau & Loke, 2021). As a result of increased parasympathetic activity and baroreflex sensitivity, a decrease in systolic and diastolic blood pressure is observed in hypertensive adults (Mourya et al., 2009). Voluntary diaphragmatic deep breathing is known to have a relaxing effect and reduce anxiety in hypertensive or prehypertensive individuals other than systolic and diastolic blood pressures (Chen et al., 2017).In the planned project, exercises, which are thought to be effective in disease management, will be created in line with the preferences of the individual and the recommendations of the physiotherapist (age, gender, BMI, etc.) and a notification will be sent when the exercise programme is created. In this way, the body mass index will remain within normal limits as the individual exercises regularly and disease management will be ensured.

In the management of hypertension, treatment compliance is also an important factor that ensures blood pressure control. As a matter of fact, the rate of blood pressure control in the world and in our country is around 25%, and the most important factor in this is non-compliance with treatment (Akan, Çaydam & Paköz, 2020). In a study conducted in our country, it was reported that 36.3% of patients complied with hypertension treatment (Akan, Çaydam & Paköz, 2020). Some of the factors that negatively affect treatment compliance are that the time allocated by the physician to the patient is not sufficient in public hospitals where the patient density is too high, and the physician-patient communication is not at the desired level, especially for individuals with chronic diseases such as diabetes, hypertension, and heart diseases (Atıcı, 2007). Significant problems that threaten patient safety may arise from lack of communication between the patient and the physician. When these patients are informed and included in the decision-making process, they are more careful about behavioural changes (such as adherence to treatment, diet, exercise). Factors such as not informing the patient about the diet to be applied during the discharge process, not explaining how to use the prescribed prescription, the physician not allocating time for informing the patient or not having time for informing the patient, and not having a suitable environment for informing in the ward negatively affect treatment compliance (Bol, Gül & Arbaycu, 2013).

ELIGIBILITY:
Inclusion Criteria:

30-65 years old Being open to communication and co-operation Having and using a smartphone Agreeing to follow a personalised diet programme Taking antihypertensive medication

Exclusion Criteria:

Illiteracy Having had MI within the last month, heart failure, valvular heart disease, exertional dyspnoea, chronic kidney disease visual problems (to be obtained from ASM records). Having a history of a disease that may cause memory impairment such as dementia, Alzheimers disease (to be obtained from ASM records).

Presence of an orthopaedic and/or neurological problem that may prevent participation in exercise

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
SF- 36 Life Quality Scale | up to three months
  The scale is a multifactor scale that includes thirty-six statements and assesses two main topics (physical and mental dimensions) and eight concepts (physical function, role limitation-physical, pain, vitality/fatigue, social function, role limitation-emotional, mental health, general health perception). A separate score is obtained for each subscale. SF-36 evaluates both negative and positive aspects of health status. The subscale scores vary between 0-100. Each health domain of the SF-36 with positive scoring in the scale is scored in such a way that the higher the score of each health domain, the higher the health-related quality of life.
Hypertension Self-Efficacy Scale | up to three months
  The scale consists of 20 items. In the original scale, the items are in 4-point Likert type ranging from "not at all appropriate" (1 point) to "very appropriate" (4 points). The total score of the scale varies between 20-80 points. An increase in the total score obtained from the scale indicates an increase in the level of self-efficacy in hypertension.

SECONDARY OUTCOMES:
International Physical Activity Scale-Short Form | up to three months
  This form, which was developed by Craig et al. to determine the physical activity levels of individuals and adapted into Turkish by Öztürk, includes 7 questions to evaluate the physical activity of individuals in the last seven days. These questions include statements to determine the sitting, walking, moderate and vigorous activities of individuals. In the calculation of the total score of this questionnaire, the MET measurements determined for sitting, walking, moderate and vigorous levels are summed and calculated. The MET value for sitting was determined as 1.5, for walking as 3.3, for moderate physical activity as 4.0 and for vigorous physical activity as 8.0. The increase in the scores obtained from the questionnaire indicates that individuals are more physically active.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers, they will be kept secret.